CLINICAL TRIAL: NCT05974397
Title: Nationwide Trends in Incidence, Healthcare Utilization, and Mortality in Hospitalized Acute Myocardial Infarction Patients in Taiwan
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BTW05
Record Dates: First submitted 2023-07-20; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- AMI: Patients with AMI
- STEMI: Patients with STEMI
- NSTEMI: Patients with NSTEMI

SUMMARY:
This was a retrospective study using the Taiwan's National Health Insurance Research Database (NHIRD). The study employed two study designs for different purposes as follows:

* A cross-sectional analysis was conducted to explore the annual incidence trends.
* A longitudinal cohort study was conducted to assess baseline characteristics, treatment patterns, long-term healthcare utilization, and cause-specific mortality among incident AMI patients.

In each part, the study was conducted for AMI, and separately for ST-segment elevation and non-ST- segment elevation myocardial infarction (STEMI and NSTEMI)

ELIGIBILITY:
Inclusion Criteria:

Cross-sectional analysis:

* Patients aged 20 years and older.
* Patients who had been admitted for AMI, defined as primary or first secondary diagnosis of AMI between 2014 and 2020.
* The diagnosis of AMI/ STEMI/ NSTEMI was identified by the International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) codes and 10th revision (ICD-10-CM) codes.
* Incident cases of AMI hospitalization were defined as no history of AMI-related hospitalization or outpatient visit within 1 year before admission.

Longitudinal analysis:

Patients aged 20 years and older.

* Patients who had been admitted for AMI, defined as primary or first secondary diagnosis of AMI between 2014 and 2017.
* The diagnosis of AMI/ STEMI/ NSTEMI was identified by ICD-9-CM codes and ICD-10-CM codes. (The ICD-9-CM code and ICD-10-CM codes were the same as above)
* Incident cases of AMI hospitalization were defined as no history of AMI-related hospitalization or outpatient visit within 1 year before admission.
* The cohort entry date was defined as the admission date of incident AMI hospitalization, and the index date was defined as the discharge date of incident hospitalization.

Exclusion Criteria:

None specified

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 124018 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Mean age of patients | 12 months
Number of male patients | 12 months
Year of patient entry into cohort | 12 months
Number of patients with AMI in Taiwan | 12 months
Number of patients with STEMI in Taiwan | 12 months
Number of patients with NSTEMI in Taiwan | 12 months
Number of AMI patients with comorbidities | Up to 3 years
Number of patients with treatment for AMI | Up to 3 years
Number of STEMI patients with comorbidities | Up to 3 years
Number of patients with treatment for STEMI | Up to 3 years
Number of NSTEMI patients with comorbidities | Up to 3 years
Number of patients with treatment for NSTEMI | Up to 3 years
Number of mortalities among AMI patients | Up to 3 years
Number of mortalities among STEMI patients | Up to 3 years
Number of mortalities among NSTEMI patients | Up to 3 years
Number of AMI patients with outpatient visits | Up to 3 years
Number of AMI patients with emergency room visits | Up to 3 years
Number of AMI patients with hospitalizations | Up to 3 years
Length of hospital stay for AMI patients | Up to 3 years
Direct medical costs for AMI patients | Up to 3 years
Number of STEMI patients with outpatient visits | Up to 3 years
Number of STEMI patients with emergency room visits | Up to 3 years
Number of STEMI patients with hospitalizations | Up to 3 years
Length of hospital stay for STEMI patients | Up to 3 years
Direct medical costs for STEMI patients | Up to 3 years
Number of NSTEMI patients with outpatient visits | Up to 3 years
Number of NSTEMI patients with emergency room visits | Up to 3 years
Number of NSTEMI patients with hospitalizations | Up to 3 years
Length of hospital stay for NSTEMI patients | Up to 3 years
Direct medical costs for NSTEMI patients | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Taipei, Taiwan